CLINICAL TRIAL: NCT06630065
Title: Translational Study of the Neural Circuits Underlying the Negative Emotional Bias of Depressive Disorders and Their Response to Ketamine
Brief Title: Study of the Neural Circuits Underlying the Negative Emotional Bias of Depressive Disorders and Their Response to Ketamine
Acronym: EMOKET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D22-P015
Record Dates: First submitted 2024-09-26; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Experimental): Depressed patients treated with Esketamin
  Interventions: Behavioral: fMRI with emotional task and pupillometry; Behavioral: Behavioral task with emotional facial expressions; Genetic: Biological investigation
- healthy volunteers (Other): Healthy subjects
  Interventions: Behavioral: fMRI with emotional task and pupillometry; Behavioral: Behavioral task with emotional facial expressions; Genetic: Biological investigation

INTERVENTIONS:
Behavioral: fMRI with emotional task and pupillometry — Anatomical and functional magnetic resonance imaging (fMRI) imaging sequences with pupillometry (~90 min)
  A functional sequence - Task (~20min):
  * Emotional task in fMRI: Instructions: simply look images, then evaluate the emotions triggered at the end of each block; rating on a valence and intensity scale and intensity (arousal) scale.
  * Experimental conditions: positive, negative and neutral
  * Paradigm: block validated image banks: IAPS, GAPED, EMOPICS, OASIS, etc. Pupillometry: In order to collect objective data on emotional bias, we will use pupillometry (or eye-tracking) during functional MRI sequences.
Behavioral: Behavioral task with emotional facial expressions — Description of the recognized emotion joy - sadness. Test to assess the hedonic value of an olfactory stimulus (10 min)
Genetic: Biological investigation — Standard biological assessment, immuno-inflammatory profile and the association of 8 mRNA editing variants

SUMMARY:
Major depressive disorder is the leading cause of disability worldwide, affecting up to 300 million people each year, and one in five people will experience depression at least once in their lives. Emotional bias is an essential component of characterized depressive episodes, leading depressed patients to attribute a more negative valence to emotional stimuli.

On the basis of recent and robust neuroscientific data revisiting the role of the cerebral amygdala as an essential essential structure for encoding the negative and positive valences and of emotional stimuli, the team has shown in mice that a depressive phenotype induced by a chronic administration of corticosterone, a well-known model of depression, is associated with a change in hedonic value allocation, i.e. pleasant odors become less pleasant, and aversive odors become even more unpleasant, mimicking what happens in humans (identical data in humans).

It assumes that:

1. There is a negative emotional bias in depressed patients compared with control subjects, evidenced by the assignment of more negative valences when viewing images.
2. In depressed subjects, compared with controls subjects, there is greater activation of the basolateral amygdala/ventral hippocampus pathway (the level of imaging resolution of imaging does not allow to study the basolateral amygdala/central amygdala pathway in humans) and less of the basolateral amygdala/nucleus accumbens pathway.
3. In depressed subjects, improvement in negative emotional bias correlated with a good response after after 4 weeks of treatment with esketamine (Spravato) measured by a 50% reduction in the Montgomery-Åsberg Depression Rating Scale.
4. In depressed patients, early improvement of emotional bias (after a single administration) is predictive of response to treatment at 4 weeks.
5. In depressed patients with a good response to a single 4-weeks course of esketamine (Spravato), a normalization of activation of basolateral amygdala/ventral hippocampus and basolateral amygdala/nucleus accumbens pathways is observed.
6. Depressed subjects have different immunoinflammatory and RNA editing patterns different from control subjects.
7. In depressed patients, clinical improvement correlates with normalization of patients; inflammatory profile and certain mRNA editing
8. Some clinical features of major depressive disorder are associated with greater negative emotional bias significant

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria :

* Age over 18
* Patient hospitalized or consulting at GHU Paris Psychiatrie et Neurosciences
* Patient with EDC (unipolar or bipolar) diagnosed according to the DSM-5 CRITERIA
* With MADRS score > 20
* For whom a course of esketamine has been decided by the psychiatrist of the patient
* Patient having given written informed consent
* Patient covered by a social security plan

Inclusion criteria for control subjects :

* Over 18 years old
* No EDC assessed by MADRS < 8

Exclusion Criteria:

Patient non-inclusion criteria:

* Psychiatric comorbidities: schizophrenic disorder or schizoaffective disorder, history of recreational use of ketamine
* Protected adults, persons under legal protection
* Contraindications to MRI, including refusal to be informed of the discovery of a clinically significant abnormality on MRI
* Pregnant or breast-feeding women
* Usual contraindications to esketamine :

  * Neurological comorbidity: epilepsy, neurodegenerative disease, cerebrovascular disease with recent history (< 3 months) of stroke or ischemic attack or transient ischemic attack
  * Cardiological co-morbidity: vascular aneurysm, ischemic heart disease with acute elements or stent within the previous 12 months, uncontrolled hypertension, heart failure, rhythm or conduction disorders on ECG
  * History of cirrhosis (or ALAT, ASAT or bilirubin greater than 2 N)
  * Severe chronic respiratory insufficiency

Exclusion criteria for control subjects:

* MADRS <8
* Contraindications to MRI, including refusal to be informed of a clinically significant clinically significant abnormality on MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Significant difference in negative emotional bias measured by an image perception task before vs. after esketamine treatment | 1 month
  Comparison of the negative emotional bias measured by an image perception task (valence) before vs. after esketamine treatment [Baseline/1 month of treatment].

SECONDARY OUTCOMES:
Measure of the blood oxygenation level with the Blood-Oxygen-Level Dependent (BOLD) signal obtained at the functional magnetic resonance imaging (fMRI) task in depressed patients and in control subjects | patients: at baseline (Day 0) and at the end-of study visit (6 weeks); control subjects: at baseline (Day 0)
  The blood oxygenation level is measured thanks to the blood-oxygen-level dependent (BOLD) signal obtained at the fMRI task. This signal will be recorded in depressed patients and control subjects at baseline (Day 0) and at the end-of-study visit (6 weeks after Day 0) only for patients.
Measure of the functional connectivity obtained at the resting-state functional magnetic resonance imaging (fMRI) in depressed patients and in control subjects | patients: at baseline (Day 0) and at the end-of study visit (6 weeks); control subjects: at baseline (Day 0)
  The basolateral amygdala/ventral hippocampus and basolateral amygdala/nucleus accumbens (BLA/vHPC, and BLA/Nac) functional connectivity obtained at the resting-state fMRI will be recorded in depressed patients and control subjects at baseline (Day 0) and at the end-of-study visit (6 weeks) only for patients
Measure of the gray matter integrity obtained at the High-resolution anatomical (T1) magnetic resonance imaging (MRI) in depressed patients and in control subjects | Patients: at baseline (Day 0) and at the end-of study visit (6 weeks); control subjects: at baseline (Day 0)
  The gray matter integrity obtained at the T1 (longitudinal relaxation time) MRI will be recorded in depressed patients and control subjects at baseline (Day 0) and at the end-of-study visit (6 weeks) only for patients
Measure of the white matter integrity obtained at the diffusion imaging in depressed patients and in control subjects | Patients: at baseline (Day 0) and at the end-of study visit (6 weeks); control subjects: at baseline (Day 0)
  The white matter integrity obtained at the diffusion imaging will be recorded in depressed patients and control subjects at baseline (Day 0) and at the end-of-study visit (6 weeks) only for patients.
Measure of the depression severity in patients and control subjects thanks to the Montgomery-Åsberg Depression Rating Scale score | Patients: at baseline (Day 0), Day 7, Week 2 (2 times), Week 3 (2 times), Week 4 (2 times), Week 5 (2 times) and at the end-of-study visit (Week 6); control subjects: at baseline (Day 0)
  The depression severity will be assessed by the investigator with the Montgomery-Åsberg Depression Rating Scale (MADRS). The depression severity score will be then calculated. Score range (min - max): 0 - 60. Higher score relates to high depression severity. The questionnaire will be realized in depressed patients and control subjects at baseline (day 0) and throughout the study only for patients.
Assessment of the emotional bias measured by an image perception task | Patients: at baseline (Day 0) and at the end-of-study visit (Week 6); control subjects: at baseline (Day 0)
  The task used to calculate the emotional bias score involves presenting images to patients and control subjects, each of which has normative ratings for valence and arousal. The objective is to present ten images per block (9 blocks repeated 3 times) allowing for an evaluation of high, neutral or low emotional valence as well as high, low or medium arousal levels. The results for each participant will be summarized in a contingency table. The total emotional bias score (accuracy score) will be calculated at baseline (Day 0) for patients and control subjects and at the end-of-study (Week 6) only for patients.
Measure of the suicidality score in depressed patients thanks to the Columbia-Suicide Severity Rating Scale | At baseline (Day 0) and at the end-of-study visit (Week 6)
  The suicidality will be assessed by the investigator with the Columbia-Suicide Severity Rating Scale. The suicidality score will be then calculated. The suicidal ideation section is rated on a scale from 1 to 5, with increasing severity from passive thoughts of death to active suicidal intent with a plan. The Suicidal Behavior section assesses past suicide attempts or preparation, with a focus on the presence and severity of suicidal actions. There is no overall score in C-SSRS but the investigator will evaluate the individual's risk level at baseline (Day 0) and at the and-of-study visit (Week 6) in depressed patients.
Measure of anhedonia score in depressed patients thanks to the Snaith-Hamilton Pleasure Scale | At baseline (Day 0) and at the end-of-study visit (Week 6)
  The Snaith-Hamilton Pleasure Scale (SHAPS) is used to measure the anhedonia. The total score ranges from 0 to 14 and is proportional to the degree of anhedonia. The questionnaire will be realized in depressed patients at baseline (day 0) and at the end-of-study visit in depressed patients.
Measure of the anxiety score in depressed patients thanks to the Beck anxiety scale | At baseline (Day 0) and at the end-of-study visit (Week 6)
  The Beck anxiety scale consists of 21 self-reported items used to assess the intensity of physical and cognitive anxiety symptoms during the past week. The total score ranges from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63). The questionnaire will be realized in depressed patients at baseline (day 0) and at the end-of-study visit in depressed patients.
Measure of the emotional reactivity in depressed patients and control subjects thanks to the Multidimensional Assessment of Thymic States scale | Patients: at baseline (Day 0), Day 7, Week 2 (2 times), Week 3 (2 times), Week 4 (2 times), Week 5 (2 times) and at the end-of-study visit (Week 6); control subjects: at baseline (Day 0).
  The MAThyS is a visual analogic scale consisting of 20 items. Score is determined line-by-line and varies from 0 to 10 for each line (centimeters). A score of 0 indicates an inhibition of the state evaluated by the item. A score of 5 indicates no change from the patient's usual state. A score of 10 corresponds to excitation for the evaluated state. An overall score between 0 and 200 is thus obtained. The questionnaire will be realized in depressed patients and control subjects at baseline (day 0) and throughout the study only for patients.
Measure of the mania score in depressed patients and control subjects thanks to the Young Mania Rating Scale | Patients: at baseline (Day 0), Day 7, Week 2 (2 times), Week 3 (2 times), Week 4 (2 times), Week 5 (2 times) and at the end-of-study visit (Week 6); control subjects: at baseline (Day 0)
  The Young Mania Rating Scale (YMRS) has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. The total score ranges from 0 to 44 and is proportional to the degree of mania. The questionnaire will be assessed by the investigator at baseline (Day 0) in patients and control subjects as well as throughout the study for patients.
Assessment of the severity and improvement of the clinical condition using the Clinical Global Impression Severity scale | Patients: at baseline (Day 0), Day 7, Week 2 (2 times), Week 3 (2 times), Week 4 (2 times), Week 5 (2 times) and at the end-of-study visit (Week 6); control subjects: at baseline (Day 0)
  The Clinical Global Impression scale (CGI) will be used by the physician to assess, with a 7-point scale, the depression severity of the patient's clinical condition, as well as, the improvement in the patient's clinical condition following treatment. Each of these scales is rated from 0 to 7. A score of 7 indicates the maximum level of severity of the patient's depressive state, and in the other case, a score of 7 indicates the maximum worsening of the patient's condition. The questionnaire will be assessed by the physician at baseline (Day 0) in patients and control subjects as well as throughout the study for patients.
Assessment of the moral pain in depressed patients with the Psychological and Physical Pain Visual Analog Scale (PPP-VAS) | At baseline (Day 0) and at the end-of-study visit (Week 6)
  Patients complete the Psychological and Physical Pain Visual Analog Scale (PPP-VAS) at baseline (Day 0) and at the end-of-study visit (Week 6). The PPP-VAS consists of six dimensions presented as paper-based visual analog scales, which patients must annotate from 0 to 10, measuring current, mean and worst pain over the last 15 days, for physical then psychological pain (0 corresponding to no pain and 10 corresponding to the maximum imaginable pain).
Assessment of the present-state dissociative symptoms score in depressed patients with the Clinician Administered Dissociative States Scale (CADSS) | At Day 7, Week 2 (2 times), Week 3 (2 times), Week 4 (2 times) and at Week 5 (2 times)
  The Clinician Administered Dissociative States Scale (CADSS) is administered by a physician to patients at Day 7, Week 2, Week 3, Week 4 and Week 5. This scale consists of 23 items, each rated from 0 to 4, with 0 indicating the absence of symptoms and 4 indicating the maximum severity of the symptom. The total score ranges from 0 (complete absence of dissociative symptoms) to a maximum score of 92 (highest level of dissociation).
Measure of the cognitive complaints score with the Cognitive complaints in Bipolar disorder Rating Assessment (COBRA) | Patients: at baseline (Day 0) and at the end-of-study visit (Week 6); control subjects: at baseline (Day 0)
  The cognitive complaints in Bipolar disorder Rating Assessment (COBRA) consists of 16 items that are rated using a 4-point scale, 0 = never, 1 = sometimes, 2 = often, and 3 = always. The COBRA total score is obtained when the scores of each item are added up (min-max score range: 0 - 48). The higher the score, the more subjective complaints. The COBRA is a self-questionnaire. Patients and control subjects will complete this questionnaire at baseline (Day 0) and patients will also complete it at the end-of-study visit (Week 6).
Assessment of the apathy score with the Starkstein Apathy Scale | At baseline (Day 0) and at the end-of-study visit (Week 6)
  The Starkstein Apathy Scale is a self-questionnaire that consists of 14 items that are rated using a 4-point scale (from 0 to 3). The total score is is obtained when scores of each item are added up (min-max score range: 0 - 42). The highest score is associated with the most significant apathy. Patients included in the current study will complete this questionnaire at baseline (Day 0) and at the end-of-study visit (Week 6).
Analysis of immune-inflammatory markers and RNA editing markers in patients and control subjects | Patients: at baseline (Day 0), Week 2, at the end-of-study visit (Week 10); control subjects: at baseline (Day 0)
  Blood samples are collected from patients at baseline (Day 0), at the second week and at the end-of-study visit (Week 6), as well as from healthy subjects at baseline (Day 0). These blood samples will allow for the analysis of immune-inflammatory markers as well as the analysis of RNA editing markers.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Henry, Pr, Principal Investigator — GHU Paris Psychiatry & Neurosciences
Locations (1):
- - Groupe hospitalo-universitaire Paris Psychiatrie et Neurosciences, Paris, Paris, France